CLINICAL TRIAL: NCT05997381
Title: REinForce: A Prospective, Single Blind, Multi-Center, Randomized, Controlled, Pivotal Study to Evaluate the Safety and Effectiveness of the BioBrace® Implant During Arthroscopic Repair of Full Thickness Rotator Cuff Tears
Brief Title: BioBrace® Implant for Arthroscopic Repair of Full Thickness Rotator Cuff Tears
Acronym: REinForce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-BB0003
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff tear; Full thickness tear; BioBrace
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BioBrace Augment Group (Experimental): An arthroscopic rotator cuff repair is performed with the BioBrace Implant fixed on top of the repaired tendon using anchors.
  Interventions: Device: Arthroscopic rotator cuff repair with BioBrace® Implant augmentation.
- Repair Only Group (Sham Comparator): An arthroscopic rotator cuff repair is performed using standard surgical procedure.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Device: Arthroscopic rotator cuff repair with BioBrace® Implant augmentation. — An arthroscopic rotator cuff repair will be performed and augmented with the BioBrace® Implant. The BioBrace® Implant is intended for use in surgical procedures for reinforcement of soft tissue where weakness exists. It is a bioresorbable, biocomposite scaffold composed of a highly porous collagen sponge and reinforced with poly-L-lactic-acid (PLLA). When used in rotator cuff repairs, it is placed on top of the tendons to augment and reinforce the underlying repair. The BioBrace® is designed to mechanically and biologically augment weakened or torn soft tissue and can be integrated into surgeons' standard of care rotator cuff repair techniques.
  Arms: BioBrace Augment Group
Procedure: Arthroscopic rotator cuff repair — An arthroscopic rotator cuff repair is performed using standard surgical procedure.
  Arms: Repair Only Group

SUMMARY:
This study aims to evaluate the safety and effectiveness of arthroscopic rotator cuff repair augmented with the BioBrace® Implant vs. arthroscopic rotator cuff repair alone in subjects requiring surgical intervention for a full-thickness rotator cuff tear.

DETAILED DESCRIPTION:
This is a prospective, single blind, multi-center, randomized, controlled, pivotal clinical study investigating the treatment of full thickness tears of the rotator cuff. Tears must involve the supraspinatus and/or infraspinatus tendons and measure ≥ 2 cm and < 5 cm. Subjects meeting the inclusion/exclusion criteria will be enrolled and will undergo either arthroscopic rotator cuff repair augmented with the BioBrace® Implant or arthroscopic rotator cuff repair alone. Clinical evaluations will be conducted at baseline (pre-operatively) and at 6 weeks, 3-, 6-, and 12-months post-operatively using various patient-reported outcome measures and MRI to assess repair integrity and re-tear rate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 40 to 70 years old
2. Positive diagnostic imaging by MRI within 6 months of enrollment of the index shoulder indicating a full thickness rotator cuff tear (RCT):

   1. Tear of the supraspinatus and/or infraspinatus tendons
   2. Tear size ≥ 2 cm and < 5 cm
3. Chronic shoulder pain ≥ 3 months
4. Failed non-operative treatment of the index shoulder to include one or all of the following:

   1. Oral analgesics
   2. Nonsteroidal anti-inflammatory medications (NSAIDs)
   3. Corticosteroid injections
   4. Activity modifications
   5. Physical therapy or home-guided exercises
5. Able to read and understand the study REB/IRB approved Informed Consent Form (ICF)
6. Willing to be available to attend each protocol-required follow-up examination

Intraoperative Inclusion Criteria:

1. Full thickness tear of the supraspinatus and/or infraspinatus tendons
2. Tear size ≥ 2 cm and < 5 cm
3. Able to reapproximate the tendons to cover > 50% of the footprint on the greater tuberosity

Exclusion Criteria:

1. Previous surgery of the index shoulder one year prior to the study surgery excluding diagnostic arthroscopy
2. Fatty infiltration of the index shoulder rotator cuff muscle ≥ Grade 3 (Goutallier Score)
3. Major medical condition that could affect quality of life and influence the results of the study as determined by the Investigator
4. Oral steroid use or steroid injection within 6 weeks prior to surgery
5. Active smoker
6. History of insulin-dependent diabetes
7. Documented evidence of a history (e.g., liver testing) of drug/alcohol abuse within 12 months of enrollment
8. Hypersensitivity to any investigational device materials including collagen of animal origin (bovine type-I), poly-L-lactic acid (PLLA) or polyethylene glycol (PEG)
9. Presence of an implanted metallic device or other implants that would contraindicate acquisition or inhibit radiologist review of an MRI of the index shoulder
10. History of claustrophobia that would prevent an MRI of the index shoulder
11. Females of child-bearing potential who are either pregnant or breastfeeding or plan to become pregnant during the course of the study
12. Currently participating, or plans to enroll in another clinical trial during this study that would affect the outcomes of this study as determined by the Investigator
13. History of non-compliance with medical treatment or clinical trial participation
14. The subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant with protocol required follow-up
15. Any comorbidity or condition that renders the patient a poor surgical candidate as determined by the Investigator
16. The subject is receiving prescription narcotic pain medication
17. The subject currently has an acute infection in the area surrounding the surgical site
18. Contralateral shoulder condition where rotator cuff repair is scheduled or to be scheduled over the course of this study
19. The subject's condition represents a worker's compensation case

Intraoperative Exclusion Criteria:

1. Subject requires subscapularis repair other than a repair with a single anchor

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
6 Month Retear Rate | 6 months post-op
  The between-group difference in radiological incidence (MRI) of a Sugaya Type IV or V full-thickness discontinuity at postoperative Month 6.

SECONDARY OUTCOMES:
12 Month Retear Rate | 12 months post-op
  The between-group difference in radiological incidence (MRI) of Sugaya Type IV or V full-thickness discontinuity at postoperative Month 12.
Single Assessment Numeric Evaluation (SANE) | Baseline, 6 weeks, 3-, 6-, and 12-months post-op
  Adjusted mean between-group difference in SANE score from baseline to 6 weeks, 3-, 6-, and 12-months post-op
Western Ontario Rotator Cuff Index (WORC) | Baseline, 6 weeks, 3-, 6-, and 12-months post-op
  Adjusted mean between-group difference in WORC score from baseline to 6 weeks, 3-, 6-, and 12-months post-op
EuroQOL Five Dimensions Questionnaire (EQ-5D-5L) | Baseline, 6 weeks, 3-, 6-, and 12-months post-op
  Adjusted mean between-group difference in health-related, quality of life from baseline to 6 weeks, 3-, 6-, and 12-months post-op

CONTACTS AND LOCATIONS:
Locations (1):
- ConMed, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No